CLINICAL TRIAL: NCT03080194
Title: The Effect of a Community-based Long-acting Antipsychotic-treated Management Model on the Violence Risk of Patients With Schizophrenia: a 1-year, Open-label Randomized Controlled Study
Brief Title: The Effect of a Community-based LAI-treated Management Model on the Violence Risk of Patients With Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maosheng Fang (Other)
Responsible Party: Sponsor-Investigator, Maosheng Fang, Research clinician, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WG17A001
Record Dates: First submitted 2017-03-02; First posted 2017-03-15 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; violence risk; long-acting antipsychotics; community-based
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- paliperidone palmitate group (Experimental): The subjects in experimental group will be injected with 150mg eq and 100mg eq paliperidone palmitate in the deltoid at the 1st and 8th day, and afterwards a flexible dose of paliperidone palmitate from 75 to 150mg eq will be administrated monthly according to clinical judgement.
  Interventions: Drug: paliperidone palmitate
- control group (Active Comparator): The subjects in control group will be applied with oral antipsychotics or other conventional medication.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: paliperidone palmitate — Subjects in experimental group will be injected with 150mg eq and 100mg eq paliperidone palmitate in the deltoid at the 1st and 8th day, and afterwards a flexible dose of paliperidone palmitate from 75 to 150mg eq will be administrated monthly according to clinical judgement. Previous oral antipsychotics could be continued or withdrawn in 2-4 weeks after first paliperidone palmitate administration according to doctors' clinical judgement.
  Other Names: Sustenna
  Arms: paliperidone palmitate group
Drug: control group — Subject in control group will be applied with oral antipsychotics or other conventional medication.
  Arms: control group

SUMMARY:
This is a 12-month open-label randomized controlled study. Patients with schizophrenia and violence risk under the government supervision will be enrolled in the study. A community-based long-acting antipsychotics-treated management model will be applied to the experimental group, which means that professional psychiatrists will provide guidance to primary-level mental health workers on the psychotic treatment, and monthly-injected long-acting antipsychotic, paliperidone palmitate, will be used in the schizophrenia treatment. Every subject in experimental group will be equipped with an intelligent robot capable at push-to-talk and push-to-view, allowing the patients and caregivers to contact doctors for assistance at any time.

The subjects in experimental group will be injected with 150mg eq and 100mg eq paliperidone palmitate in the deltoid at the 1st and 8th day, and afterwards a flexible dose of paliperidone palmitate from 75 to 150mg eq will be administrated monthly according to clinical judgement.

Subjects in control group will be treated with oral antipsychotics or other conventional medication.

DETAILED DESCRIPTION:
This is a 12-month open-label randomized controlled study. Patients with schizophrenia and violence risk under the government supervision will be enrolled in the study. A community-based long-acting antipsychotics-treated management model will be applied to the experimental group, which means that professional psychiatrists will provide guidance to primary-level mental health workers on the psychotic treatment, and monthly-injected long-acting antipsychotic, paliperidone palmitate, will be used in the schizophrenia treatment. Every subject in experimental group will be equipped with an intelligent robot capable at push-to-talk and push-to-view, allowing the patients and caregivers to contact doctors for assistance at any time, if they are able to use smart phones.

The subjects in experimental group will be injected with 150mg eq and 100mg eq paliperidone palmitate in the deltoid at the 1st and 8th day, and afterwards a flexible dose of paliperidone palmitate from 75 to 150mg eq will be administrated monthly according to clinical judgement. Previous oral antipsychotics could be continued or withdrawn in 2-4 weeks after first paliperidone palmitate administration according to doctors' clinical judgement. Doctors have rights to decide whether a patient needs in-hospital treatment or extramural hospital treatment. The study protocol does not limit other medication or treatment measures except the injectable paliperidone palmitate. Other medication or treatment measures should be decided according to doctors' clinical judgement and negotiation with patients and guardians.

Subjects in control group will be treated with oral antipsychotics or other conventional medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders , Fifth Edition (DSM-V) and rated under 70 in PANSS;
* Had violent behavior such as smashing or breaking, threatening with a weapon, commiting arson or explosion in the past one year, whether the behavior can be stopped by persuading or not;
* Living with a guardian or a caregiver;
* Informed consent from the patients or their guardians;
* Resulted negative in urine pregnancy test if female at their reproductive age; female subjects must take effective measures to prevent pregnancy during the whole study or have been postmenopausal.

Exclusion Criteria:

* Patients who have had suicidal ideation or suicidal attempts within 12 months before screening or in screening period;
* Intravenous drug abuse or Opioid dependence within 3 months before screening;
* Patients with treatment-resistant schizophrenia;
* Large dose of Clozapine (≥200mg/day) or other long-acting injectable antipsychotics used within 3 months or within 2 drug half-life periods before screening;
* Patients with any severe or unstable cardiovascular, respiratory, nervous system or other system diseases; clinically significant abnormality in laboratory examinations or ECG;
* Communication difficulties caused by cognitive impairment or unable to complete the assessments in the study;
* Patients assessed as unsuitable for the study in other reasons, such as allergic or intolerant to risperidone or paliperidone, resistant to risperidone or paliperidone (ineffective after adequate dosage and duration in medical history); unable to provide informed consent; historical treatments which might effect the results of the study; historical neuroleptic malignant syndrome or tardive dyskinesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Violence Risk Assessment For Severe Psychiatric Patients | 1 year
  The percentage of subjects rated as no or low risk (scored 0 or 1) in Violence Risk Assessment For Severe Psychiatric Patients after 1-year treatment

SECONDARY OUTCOMES:
Modified Overt Aggression Scale (MOAS) | 1 year
  Patients' rated score in Modified Overt Aggression Scale after 1-year treatment
Health economic evaluation | 1 year
  The patients' and the caregivers' health economic questionnaire after 1-year treatment
Positive and Negative Syndrome Scale (PANSS) | 1 year
  PANSS total score after 6-month and 1-year treatment
Hospitalization frequency | 1 year
  Hospitalization frequency after 6-month and 1-year treatment
WHO Quality of Life-BREF (WHOQOL-BREF) | 1 year
  The patients' and the caregivers' WHOQOL-BREF score after 6-month and 1-year treatment
Visual Analogue Scale-100 (VAS 100) | 1 year
  The patients' and the caregivers' VAS 100 score after 6-month and 1-year treatment
Family Burden Scale of Diseases (FBS) | 1 year
  Family burden of the patient's family
Personal and Social Performance Scale (PSP) | 1 year
  PSP global score after 6-month and 1-year treatment
Treatment Emergent Symptom Scale (TESS) | 1 year
  Treatment Emergent Symptom Scale (TESS) score after 6-month and 1-year treatment
Vital signs | 1 year
  Heart rate and blood pressure after 6-month and 1-year treatment
Clinical laboratory examination | 1 year
  Blood routine examination after 6-month and 1-year treatment
Electrocardiogram (ECG) | 1 year
  Electrocardiogram (ECG) after 6-month and 1-year treatment
Adverse events | 1 year
  The frequency of adverse events in the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lee, Doctor, Study Director — Wuhan Mental Health Centre

IPD SHARING:
Plan to Share IPD: Undecided